CLINICAL TRIAL: NCT05875987
Title: Pilot Study Evaluating the Clinical Performance of the Quantra With the QStat Cartridge at the Point-of-care in Obstetric Patients
Brief Title: Evaluation of the Quantra QStat System in Obstetric Patients
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-044
Record Dates: First submitted 2023-04-28; First posted 2023-05-25 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Blood Loss Massive; Post Operative Hemorrhage
Keywords: Quantra; Viscoelastic testing; Coagulation
MeSH Terms: conditions — Postoperative Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Obstetric Patients: Obstetric patient population experiencing excessive bleeding around the time of delivery
  Interventions: Device: Quantra System

INTERVENTIONS:
Device: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: QStat Cartridge

SUMMARY:
This pilot study will assess the performance of the Quantra System with the QStat Cartridge versus standard of care coagulation testing in bleeding pregnant women at delivery.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The QStat Cartridge was developed to monitor hemostasis in patients that may experience a range of coagulopathies of various etiologies including fibrinolytic defects. These patients include the tobstetric hemorrhage population. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed in parallel yielding five parameters that depict the functional status of a patient's coagulation system.

This single-center, prospective, observational pilot study will evaluate the performance of the Quantra System with the QStat Cartridge as compared to standard of care coagulation testing in bleeding pregnant women at delivery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years.
* Subject is pregnant or at least 24 h postpartum
* Subject is fluent in English language.
* Subject is experiencing significant bleeding resulting in activation of the stage 2 OB hemorrhage protocol as defined by blood loss ≥1500ml at delivery or within the first 24 hours after delivery, and/or is hemodynamically unstable and/or is experiencing increased abnormal bleeding not responsive to OB stage 1 hemorrhage resuscitation.
* Subject or subject's legally authorized representative (LAR) is willing to provide informed consent, either prospectively or by deferred consent.

Exclusion Criteria:

* Subject is incarcerated at the time of the study.
* Subject is currently enrolled in a distinct study that might confound the results of the proposed study
* Subject is affected by a condition that, in the opinion of the clinical team, may pose additional risks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females
Study Population: Pparturients 18 years or older who experience an obstetric hemorrhage around the time of delivery or cumulatively over 24h after delivery or unstable vital signs or clinical signs of a coagulopathy managed with activation of the stage 2 OB hemorrhage protocol.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time to laboratory aPTT test results | At the time the OB hemorrhage protocol is activated, anticipated with 24 hours after birth
  Coagulation function assessed by Quantra Clot Time (CT, sec) and activated partial thromboplastin (aPTT, sec) test
Comparison of Quantra Fibrinogen Contribution to Clot Stiffness to laboratory coagulation fibrinogen test results | At the time the OB hemorrhage protocol is activated, anticipated with 24 hours after birth
  Coagulation function assessed by Quantra Fibrinogen Contribution to Clot Stiffness (FCS, hPa) and Clauss fibrinogen (mg/dL) test
Comparison of Quantra Clot Time to ROTEM delta INTEM CT test results | At the time the OB hemorrhage protocol is activated, anticipated with 24 hours after birth
  Coagulation function assessed by Quantra Clot Time (CT, sec) and ROTEM INTEM CT (sec) test
Comparison of Quantra Fibrinogen Contribution to Clot Stiffness to ROTEM delta FIBTEM test results | At the time the OB hemorrhage protocol is activated, anticipated with 24 hours after birth
  Coagulation function assessed by Quantra Fibrinogen Contribution to Clot Stiffness (FCS, hPa) and ROTEM FIBTEM (mm) test

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No